CLINICAL TRIAL: NCT06267209
Title: Conditioned Pain Modulation in Patients With Hemophilic Arthropathy. A Cross-sectional Cohort Study
Brief Title: Conditioned Pain Modulation in Patients With Hemophilia
Status: Recruiting | Type: Observational
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Other Study IDs: He-Modulation
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia
Keywords: Haemophilia; Joint pain; Conditioned pain modulation; Kinesiophobia; Catastrophism; Anxiety
MeSH Terms: conditions — Hemophilia A; Arthralgia; Kinesiophobia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observacional group: Patients will be recruited in 3 regions of Spain (Galicia, Madrid and Malaga), through the respective provincial associations and the Spanish Federation of Hemophilia.
  The assessment will take place at the premises of the hemophilia associations included in the study. All the evaluations will be carried out by the same physiotherapist, following the same evaluation protocol.
  The primary variable of the study will be the conditioned modulation of pain, being age the dependent variable. Secondary variables, estimated as modifiers or confounders, will be kinesiophobia, catastrophizing, anxiety perception, joint damage, pain intensity, functional capacity and pain threshold to pressure, and type of treatment and development of inhibitors.
  Interventions: Other: Observational group

INTERVENTIONS:
Other: Observational group — After confirming that the patients not meet any of the exclusion criteria, dependent and confounding study variables will be assessed.
  Patients will be recruited in 3 regions of Spain (Galicia, Madrid and Malaga), through the respective provincial associations and the Spanish Federation of Hemophilia.
  The assessment will take place at the premises of the hemophilia associations included in the study. All the evaluations will be carried out by the same physiotherapist, following the same evaluation protocol.
  The primary variable of the study will be the conditioned modulation of pain, being age the dependent variable. Secondary variables, estimated as modifiers or confounders, will be kinesiophobia, catastrophizing, anxiety perception, joint damage, pain intensity, functional capacity and pain threshold to pressure, and type of treatment and development of inhibitors.

SUMMARY:
Introduction: Hemophilic arthropathy is characterized by functional alterations, disabling physical sequelae, and chronic pain. Conditioned pain modulation describes the net effect of endogenous pathways that enhance or diminish the effects of afferent noxious stimuli.

Objectives: To describe conditioned pain modulation in patients with hemophilia and identify the best predictive model of conditioned pain modulation in these patients Methods: Cross-sectional cohort study. 51 patients with hemophilic arthropathy will be recruited in 3 regions of Spain. The main study variable will be the conditional pain modulation (Conditioned Pain Modulation Index, using an ischemic technique of the arm using the pain pressure threshold as a test stimulus), with age being the dependent variable. The secondary variables, estimated as modifying or confounding variables, will be kinesiophobia (Tampa Scale for Kinesiophobia), catastrophizing (Pain Catstrophizing Scale), trait and state anxiety (State-Trait Anxiety Inventory) and the main clinical, anthropometric, and sociodemographic.

Expected results: Identify the degree of modulation conditioned by pain in patients with hemophilic arthropathy. Identify the best predictive model for conditioned pain modulation in these patients based on the study variables

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A or B.
* Patients over 18 years of age.
* Persons with a medical diagnosis of bilateral hemophilic ankle arthropathy.
* Patients with clinical assessment by Hemophilia Joint Health Score (>4 points).
* Persons with hemophilia on prophylactic treatment with FVIII / FIX coagulation concentrates or monoclonal antibodies.
* Have signed the informed consent document.

Exclusion Criteria:

* Patients with neurological or cognitive alterations that prevent the comprehension of the questionnaires and physical tests.
* Patients who have had an ankle hemarthrosis in the 6 months prior to the start of the study.
* Patients who have taken analgesic or anti-inflammatory drugs in the 30 days prior to the study.
* Patients who are undergoing an intervention (physiotherapeutic or orthopedic) at the time of the study.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 51 patients with hemophilic ankle arthropathy has been estimated.
  The assessment will take place at the premises of the hemophilia Associations included in the study. All evaluations will be performed by the same physical therapist, following the same evaluation protocol.
  Given the characteristics of the study, the risks of bleeding in these patients during the evaluations should be minimized by designing a well-structured and justified protocol. Likewise, it should be emphasized that the study does not imply any change in the routines and medical management guidelines of the patient with respect to the usual clinical follow-up conditions, following the premises of the physician who usually attends the patient at his or her referral hospital.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-03 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Assess the Conditioned Pain Modulation Index | Screening visit
  First, we will measure the pain threshold to pressure at the base of the dorsal part of the distal phalanx of the thumb, and then we will provoke the conditioned stimulus using the ischemia test on the contralateral upper limb. For the ischemia test, a sphygmomanometer will be used and inflated to 240 mmHg. The arm will be positioned horizontally. Patients will be asked to indicate the intensity of pain on a numerical pain rating scale until a pain rating of 7/10 appears. Patients will perform resistance exercises in wrist extension by lifting a 2 kg weight up to a maximum of 45 repetitions. With the sphygmomanometer still inflated, pain detection threshold measurements will be repeated at the dorsal aspect of the distal phalanx of the thumb. The time shall not be extended beyond six minutes.

SECONDARY OUTCOMES:
Assess the kinesiophobia with Tampa Scale of Kinesiophofia | Screening visit
  With the Tampa Scale of kinesiophobia (TSK-11SV) questionnaire, the fear of movement of the patients included in the study will be evaluated. It consists of 11 items. Its values have a range of 1 to 4 points, where the higher the score, the greater the fear of movement
Assess the catastrophizing with Pain catastrophizing scale | Screening visit
  With the Pain catastrophizing scale questionnaire, the catastrophizing of patients with congenital coagulopathies will be measured. The scale, made up of 13 items, is assessed with a range of 0 to 4 points (lower score indicates less catastrophism).
Assess the catastrophizing with State-Trait Anxiety Inventory | Screening visit
  With the State-Trait Anxiety Inventory (STAI) scale, the perception of anxiety of the patients included in the study will be measured. The state and the anxiety trait of each subject are evaluated with a score of 0 to 30 points for each scale, where a higher score indicates a higher anxiety index in the trait or state.
Assess the joint damage with Haemophilia Joint Health Score | Screening visit
  With the Hemophilia Joint Health Score scale, specific for its use in patients with hemophilia, the joint status of patients with hemophilic arthropathy will be evaluated. It evaluates 8 items: inflammation and duration of this, pain, muscle atrophy and strength, crackles, and loss of flexion and extension. It has a score of 0 (no joint damage) to 20 points (maximum joint damage) per joint (elbows, knees and ankles). A gait rating is added to the 120 points (range 0-4 points), the maximum rating on this scale being 124 points
Assess the joint pain with visual analog scale | Screening visit
  The visual analog scale will be used to assess the perception of joint pain, being valued with a range of 0 to 10 points (from no pain to the maximum pain suffered or imaginable) in the joints evaluated
Assess the pressure pain threshold with pressure algometer | Screening visit
  With a pressure algometer (model Wagner FPN100) we will measure the pressure pain threshold, at the joint level and at a distance (in another part of the body). This device measures in Newton / cm2 the pressure at which the subject perceives pain under pressure. A pressure will be made on the chosen point, which we will increase at an approximate speed of 50kPa / s until the patient warns us that the sensation begins to be painful. We will be assessed in ankle (lateral malleolus, L5 spinous process, and extensor carpi longus muscle).
Assess the functional capacity with the 6-Minute Walking test | Screening visit
  The 6-Minute Walking test is performance-based, measuring walking speed and submaximal exercise capacity. Patients are instructed to walk a 30 to 50 meter track for 6 minutes and try to cover as much distance as possible without running. The distance covered, in meters, in 6 minutes is recorded, allowing the use of a walking aid or orthosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No